CLINICAL TRIAL: NCT03393468
Title: An Open Label Randomized Phase 1 Pharmacokinetic Study of Dapivirine Gel Administered Rectally to HIV-1 Seronegative Adults
Brief Title: Pharmacokinetic Study of Dapivirine Gel Administered Rectally to HIV-1 Seronegative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTN-033; 12065 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A: Dapivirine gel (Experimental): Participants will receive 2.5 g of dapivirine gel administered rectally via an applicator, followed by a 2- to 4-week washout period. Participants will then receive a second dose of up to 10 g of dapivirine gel administered rectally via a coital simulation device.
  Interventions: Drug: Dapivirine gel
- Sequence B: Dapivirine gel (Experimental): Participants will receive up to 10 g of dapivirine gel administered rectally via a coital simulation device, followed by a 2- to 4-week washout period. Participants will then receive a second dose of 2.5 g of dapivirine gel administered rectally via an applicator.
  Interventions: Drug: Dapivirine gel

INTERVENTIONS:
Drug: Dapivirine gel — Dapivirine gel (0.05%); administered rectally

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of dapivirine gel administered rectally to HIV-1 seronegative adults.

DETAILED DESCRIPTION:
This study will evaluate the pharmacokinetics (PK) of dapivirine gel administered rectally to HIV-1 seronegative adults.

Participants will be randomly assigned to two groups: Sequence A or Sequence B. Participants in Sequence A will receive 2.5 g of dapivirine gel administered rectally via an applicator, followed by a 2- to 4-week washout period. Participants will then receive a second dose of up to 10 g of dapivirine gel administered rectally via a coital simulation device. Participants in Sequence B will receive up to 10 g of dapivirine gel administered rectally via a coital simulation device, followed by a 2- to 4-week washout period. Participants will then receive a second dose of 2.5 g of dapivirine gel administered rectally via an applicator.

Participants will be in the study for approximately 1 month and will attend 7 study visits. Study visits may include behavioral assessments, physical examinations, blood and urine collection, throat and anorectal sample collection, and PK sampling.

ELIGIBILITY:
Inclusion Criteria:

* Men and transgender women who are 18 years or older at Screening, verified per site standard operating procedure (SOP)
* Able and willing to provide written informed consent
* HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in Appendix II of the study protocol and willing to receive HIV test results
* Able and willing to provide adequate locator information, as defined in site SOP
* Available to return for all study visits and willing to comply with study participation requirements
* In general good health at Screening and Enrollment, as determined by the site Investigator of Record (IoR) or designee
* At Screening, history of consensual receptive anal intercourse (RAI) at least once in the past year per participant report
* Willing not to take part in other research studies involving drugs, medical devices, genital or rectal products, or vaccines for the duration of study participation (including the time between Screening and Enrollment)
* Willing to abstain from RAI, receptive oral anal stimulation (i.e., rimming), rectal stimulation via fingers, as well as the insertion of any non-study products into the rectum for 72 hours before and after each study visit

Exclusion Criteria:

* At Screening:

  * Hemoglobin Grade 1 or higher*
  * Platelet count Grade 1 or higher*
  * White blood count Grade 2 or higher*
  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher*
  * Serum creatinine greater than 1.3 times the site laboratory upper limit of normal (ULN)
  * International normalized ratio (INR) greater than 1.5 times the site laboratory ULN
  * Positive for hepatitis C antibody
  * Positive for hepatitis B surface antigen
  * History of inflammatory bowel disease by participant report
  * (*As per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017)
  * Note: Otherwise eligible participants with an exclusionary test result (other than HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV)) can be re-tested during the screening process. If a participant is re-tested and a non-exclusionary result is documented within 30 days of providing informed consent for screening, the participant may be enrolled.
* Known adverse reaction to latex or polyurethane (ever)
* Anticipated use of and/or unwillingness to abstain from the following medications during study participation:

  * Anticoagulant medications
  * Aspirin (greater than 81 mg/day)
  * Non-steroidal anti-inflammatory drugs (NSAIDS)
  * Any other drugs that are associated with increased likelihood of bleeding
  * Rectally-administered medications or products containing nonoxynol-9 (N-9) or corticosteroids
  * CYP3A inducer(s) and/or inhibitor(s) as specified in the MTN-033 Study Specific Procedures (SSP) Manual
  * Hormone-replacement therapy in tablet, patch, injectable or gel form
* Known adverse reaction to any of the components of the study product, applicator or coital simulation device
* Use of pre-exposure prophylaxis (PrEP) for HIV prevention within 1 month prior to Enrollment, and/or anticipated use and/or unwillingness to abstain from PrEP during trial participation
* Use of post-exposure prophylaxis (PEP) for potential HIV exposure within the 6 months prior to Enrollment
* Use of systemic immunomodulatory medications within the 6 months prior to Enrollment, and/or anticipated use during trial participation
* RAI without a condom and/or penile-vaginal intercourse with a partner who is known to be HIV-positive in the 6 months prior to Enrollment
* Non-therapeutic injection drug use in the 12 months prior to Enrollment
* Participation in research studies involving drugs, medical devices, genital or rectal products, or vaccines within 30 days of the Enrollment Visit
* Per participant report at Screening, treatment of an anogenital sexually transmitted infection (STI) (after diagnosis) within the past 3 months
* At Screening, participant-reported symptoms, and/or clinical or laboratory diagnosis of active anorectal or reproductive tract infection (RTI) requiring treatment per current CDC guidelines (http://www.cdc.gov/std/treatment) or symptomatic urinary tract infection (UTI). Infections requiring treatment include symptomatic Neisseria gonorrhea (GC), Chlamydia trachomatis (CT) infection, syphilis, active herpes simplex virus (HSV) lesions, anogenital sores or ulcers, or symptomatic genital warts, chancroid, trichomoniasis.

  * Note: Otherwise eligible participants with an exclusionary UTI may be re-tested during the screening process.
* At Enrollment, active anorectal infection or RTI requiring treatment per current CDC guidelines (http://www.cdc.gov/std/treatment) or symptomatic UTI. Infections requiring treatment include symptomatic GC, CT, syphilis, active HSV lesions, anogenital sores or ulcers, symptomatic genital warts, trichomoniasis, chancroid.

  * Note: HSV-1 or HSV-2 seropositive diagnosis with no active lesions is permitted since treatment is not required.
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Measurement of dapivirine concentrations in rectal fluid | Measured through approximately 1 month
  As assessed by pharmacokinetic sampling and analysis
Measurement of dapivirine concentrations in plasma | Measured through approximately 1 month
  As assessed by pharmacokinetic sampling and analysis
Measurement of dapivirine concentrations in rectal mucosal tissue homogenates | Measured through approximately 1 month
  As assessed by pharmacokinetic sampling and analysis

SECONDARY OUTCOMES:
Frequency of Grade 2 or higher adverse events (AEs) | Measured through approximately 1 month
  As defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 2 and 3 (Male Genital [Dated November 2007] and Rectal [Clarification Dated May 2012] Grading Tables for Use in Microbicide Studies)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Ho, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh CRS, Pittsburgh, Pennsylvania, United States